CLINICAL TRIAL: NCT03212963
Title: An Open Label Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of Twice Daily Halobetasol Propionate Lotion, 0.05% in Subjects 12 to 16 Years 11 Months of Age With Plaque Psoriasis Receiving Two Weeks of Treatment
Brief Title: Evaluation of Adrenal Suppression Potential and Pharmacokinetics of Halobetasol Lotion 0.05%
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 177-0551-201
Record Dates: First submitted 2017-04-18; First posted 2017-07-11 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Open label study to evaluate adrenal suppression potential and pharmacokinetics of halobetasol lotion 0.05%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Halobetasol lotion treatment arm (Experimental): All subjects will receive Halobetasol Topical Lotion, 0.05%.
  Interventions: Drug: Halobetasol Topical Lotion

INTERVENTIONS:
Drug: Halobetasol Topical Lotion — Halobetasol Lotion 0.05%, applied twice daily in subjects aged 12 to 16 years 11 months with stable plaque psoriasis.
  Other Names: Halobetasol topical lotion 0.05%

SUMMARY:
The objective of this open-label multicentric study is to determine the adrenal suppression potential and the pharmacokinetic (PK) properties of halobetasol lotion (HBP) applied twice daily for up to two weeks in subjects aged 12 to 16 years 11 months with stable plaque psoriasis. Subject enrollment will continue until at least 20 subjects with both screening and end of study (EOS) serum cortisol data (pre- and pos-tcosyntropin stimulation) have completed the study without any significant protocol violations (evaluable subjects). This may require the enrollment of approximately 25 subjects.

DETAILED DESCRIPTION:
This is an open label, multicenter study of an investigational formulation of HBP Lotion, 0.05% in male and female subjects aged 12 to 16 years 11 months with stable plaque psoriasis. Approximately 25 subjects with stable plaque psoriasis on at least 10% of their BSA (excluding the face, scalp, groin, axillae and other intertriginous areas), who fulfill the inclusion/exclusion criteria will be enrolled at multiple study sites. All subjects will have a screening CST to assess their HPA axis response at Visit 1 (Screening Visit).

Enrollment into the treatment phase of the study should be timed such that the screening CST will be performed a minimum of 20 days before Baseline Visit. At Visit 2 (Baseline), eligible subjects with normal adrenal function will be eligible to participate in the study.

Subjects will apply HBP Lotion, 0.05% to all psoriasis plaques identified at Visit 2 twice daily (approximately every 12 hours) for the assigned treatment period or until the investigator verifies the subject's psoriasis has cleared. The study is designed to determine the adrenal suppression potential and pharmacokinetic properties of the test article after the subject applies a maximum of approximately 50 grams per week for up to a two week treatment period. All subjects will have a CST to reassess their HPA axis response at EOS (or earlier if the investigator verifies the subject's psoriasis has cleared). In this study, an abnormal Hypothalamujs Pituitary Adrenal axis response to 0.25 milligram dose of cosyntropin is defined as a post-CST serum total cortisol level of less than equal to18 μg/dL.

Eligible subjects will have blood drawn at Screening for baseline drug concentration in plasma. On Day 8, all subjects, regardless of lesion clearance, will have blood drawn for assessment of trough drug concentration in plasma. At the Day 15 visit, subjects who have continued to treat lesions will have a final PK blood sample collected approximately 12 hours after their Day 14 evening application and just prior to the initiation of the CST.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female and is 12 to 16 years 11 months of age.
2. Subject has provided written informed assent and was accompanied by the parent or legal guardian at the time of assent/consent signing. The parent or legal guardian has provided informed consent for the subject. 3. Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 10% body surface area (BSA) within the Treatment Area. The "Treatment Area" is defined as the entire body exclusive of the face, scalp, groin, axillae, and other intertriginous areas.

4. Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit.

5. Subject is willing and able to apply the test article as directed, comply with study instructions and commit to all follow-up visits for the duration of the study.

6. Females must have a negative urine pregnancy test (UPT) at the Screening and Baseline Visits and agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
3. Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, adrenal axis function (e.g., Addison's Disease, Cushing's Syndrome) or which exposes the subject to an unacceptable risk by study participation.
4. Subject has used any phototherapy (including laser), photochemotherapy or systemic psoriasis therapy including methotrexate, retinoids, cyclosporine or biologics within 30 days prior to the initiation of treatment with the test article.
5. Subject has used systemic corticosteroids (including oral or intramuscular) or topical, inhaled or intranasal corticosteroids within 30 or 14 days, respectively, prior to Part B of the Screening Visit and/or the subject has used systemic or topical corticosteroids between Part B of the Screening Visit and the initiation of treatment.
6. Subject has had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the initiation of treatment or is intending to have such exposure during the study that is thought by the investigator to likely modify the subject's disease.
7. Subject has used topical psoriatic therapy including tar, anthralin, retinoids, vitamin D analogs (e.g., Dovonex®) within 14 days prior to the initiation of treatment with the test article.
8. Subject has used emollients/moisturizers on areas to be treated within one day prior to the initiation of treatment with the test article.
9. Subject is currently using lithium or Plaquenil (hydroxychloroquine).
10. Subject is currently using a beta-blocking medication (e.g., propranolol) or angiotensin converting enzyme (ACE) inhibitors (e.g., lisinopril) at a dose that has not been stabilized, in the opinion of the investigator.
11. Subject has a history of sensitivity to any of the ingredients in the test article.
12. Subject is pregnant, lactating, or is planning to become pregnant during the study.
13. Subject is currently enrolled in an investigational drug or device study.
14. Subject has used an investigational drug or investigational device treatment within 30 days prior to Visit 1 (Screening).
15. Subject has been previously enrolled in this study and treated with the test article.
16. Subject has an irregular sleep schedule or works night shifts (cortisol levels exhibit physiological diurnal variation).
17. Subject has a screening Cosyntropin Stimulation Test (CST) with a post 30-minute stimulation cortisol level of less than equal to 18 μg/dL.
18. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Magajna, MS, Study Chair — Therapeutics, Inc.
Locations (3):
- United States (3):
  - First OC Dermatology, Fountain Valley, California
  - Power MD Clinical Research Institute, Hialeah, Florida
  - MediSearch Clinical Trials, Saint Joseph, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Halobetasol Lotion Treatment Arm
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: safety population
Arm/Group | Halobetasol Lotion Treatment Arm
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment
Description: The IGA score (5-point scale of 0 to 4: 0[clear]; 1[almost clear]; 2[mild]; 3[moderate]; 4[severe]) is an evaluation of the overall severity of a subject's psoriasis in the Treatment Area and takes into consideration the 3 individual characteristics of psoriasis (scaling, erythema, and plaque elevation).
Time Frame: Day 15
Measure: Number; unit: number of subjects
Arm/Group | Halobetasol Lotion Treatment Arm
Number analyzed (Participants) | 14
number of subjects
  IGA Grade 0 | 5
  IGA Grade 1 | 3
  IGA Grade 2 | 4
  IGA Grade 3 | 2
  IGA Grade 4 | 0

2. Primary Outcome: Percent BSA Affected With Disease
Description: The Percent Body Surface Area (BSA) Affected with Disease was defined as the BSA which was affected with psoriasis within the Treatment Area.
Time Frame: Day 15
Population: Evaluable Population
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Halobetasol Lotion Treatment Arm
Number analyzed (Participants) | 14
percentage of body surface area | 2.8 (3.04)

3. Primary Outcome: Percent Body Surface Area Treated With Test Article
Description: The Percent Body Surface Area Treated with Test Article was defined as the BSA which was affected with psoriasis within the Treatment Area that was treated.
Time Frame: Day 8
Population: Evaluable Population
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Halobetasol Lotion Treatment Arm
Number analyzed (Participants) | 14
percentage of body surface area | 7.1 (1.98)

4. Primary Outcome: Number of Subjects With Abnormal Hypothalamus-Pituitary-Adrenal Axis Response
Description: An abnormal Hypothalamus-Pituitary-Adrenal (HPA) axis was response was defined as a 30-minute post-stimulation serum cortisol level of ≤18 μg/dL at end of study (EOS)
Time Frame: Day 15
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: number of subjects
Arm/Group | Halobetasol Lotion Treatment Arm
Number analyzed (Participants) | 14
number of subjects | 1 [0.2 to 33.9]

ADVERSE EVENTS:
Time Frame: Day 15
Arm/Group | Halobetasol Lotion Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Halobetasol Lotion Treatment Arm (N=16)
ACTH stimulation test abnormal (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03212963/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03212963/SAP_001.pdf